CLINICAL TRIAL: NCT03293199
Title: Randomized Controlled Trial on Comparison of Chest Tube Drainage and Needle Aspiration in Treatment of Spontaneous Pneumothorax
Brief Title: Comparing Efficacy of Chest Tube Drainage and Needle Aspiration in Pneumothorax Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tabriz University of Medical Sciences (Other)
Collaborators: AJA University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Ramouz, Doctor, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.AJAUMS.REC.1396.24
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Pneumothorax Spontaneous Primary; Pneumothorax, Recurrent; Pneumothorax Spontaneous Tension; Pneumothorax, Spontaneous
MeSH Terms: conditions — Pneumothorax; Recurrence

STUDY DESIGN:
Intervention Model Description: Patients will be randomly and equally assigned to study groups, as follows: group (a) will undergo chest tube drainage implementation and group (b) will undergo repetitive needle aspiration till pnuemothorax resolution.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since patients are alert and conscious, therefore we are unable to blind the participants. However, care provider will not take part in the data acquisition and outcome analysis. The investigator and outcome assessor will be blinded to patients allocated group and treatment type provided in each patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chest tube drainage (Active Comparator): This group will undergo chest tube drainage as an intervention for spontaneous pneumothorax treatment.
  Interventions: Procedure: Chest tube drainage
- Needle aspiration (Active Comparator): This group will undergo repetitive needle aspiration as an intervention for spontaneous pneumothorax treatment.
  Interventions: Procedure: Repetitive needle aspiration

INTERVENTIONS:
Procedure: Chest tube drainage — In this group, in the supine position and subsequent to prepping and draping and local anesthesia administration via lidocaine 2%, F16 or F20 (based on patients physical status) sterile plastic tube will be implemented at the level 4th or 5th intercostal space through the midaxillary line. Subsequently, the external end of the tube will be connected to water sealing bottle and water bubbles coming out will be considered as proper chest tube insertion.
  Arms: Chest tube drainage
Procedure: Repetitive needle aspiration — In this group, prior to needle aspiration, patients will take the semi-supine position. Subsequent to local anesthesia via lidocaine 2%, as well as prepping and draping, G16 intravenous angiocath will be inserted through midclavicular line at the level 2nd or 3rd intercostal space. Air bubble inside the lidocaine syringe will be considered as needled entrance to pleural cavity, thus 5-10 cm of the angiocath will be import to inside of the cavity. The catheter needle will be removed and catheter will be fixed using sterile sticks. A three-way valve will be connected to external end of the catheter and a 50 ml syringe will be connected to the valve. The air suction will be performed using 50 ml syringe till end of the air suction or up to 3.5 liters of air suctioning.
  Arms: Needle aspiration

SUMMARY:
Spontaneous pneumothorax is a common condition which is defined as air presence inside of pleural space. Despite, several studies that have been carried on management patients suffering spontaneous pneumothorax, the first step approach on patients is still the topic of debate. Since chest tube drainage and needle aspiration are widely used first step techniques in spontaneous pneumothorax, current study compares the efficacy of abovementioned techniques, as well as long-term outcomes. In current multi-center single-blinded RCT, all patients admitted with spontaneous pneumothorax will be enrolled study and written consent form provided by patients, simultaneously. Patients randomly assigned to study groups including (A) chest tube drainage and (B) needle aspiration. Subsequently, all patients will undergo one-year follow-up and will be evaluated in terms of treatment success rate and pneumothorax recurrence. Hypothesis of present trial are as follows: a) repetitive needle aspiration may lead to higher treatment success rate in patients with primary spontaneous pneumothorax, in comparison to chest tube drainage, b) needle aspiration may result in reduction of hospital admission duration in patients with primary spontaneous pneumothorax compared to chest tube drainage, c) the rate of spontaneous pneumothorax recurrence during one-year follow up might be lower in patients who undergo needle aspiration instead of chest tube drainage.

DETAILED DESCRIPTION:
The chest tube drainage and needle aspiration are widely used first step techniques in spontaneous pneumothorax, thus present randomized controlled trial (RCT) aims to compare the efficacy of abovementioned techniques, as well as long-term outcomes. The study protocol has been confirmed by the ethics committee of AJA University. In current multi-center single-blinded RCT, all patients admitted with primary spontaneous pneumothorax will be enrolled study and written consent form provided by patients, simultaneously. With due attention to the success rate of 18% provided in a previous study comparing primary spontaneous pneumothorax treatment procedures and the study power of 80% and the confidence coefficient of 0.05, study population calculated to include 64 patient, which increased to 70 patients with taking 10% of falling risk into consideration. Using Randlist software, patients will be randomly assigned to study groups including (A) chest tube drainage and (B) needle aspiration. Subsequently, all patients will undergo one-year follow-up and will be evaluated in terms of treatment success rate and pneumothorax recurrence.

In chest tube drainage group, while the patient is positioned in the supine position and subsequent to local anesthesia administration via lidocaine 2%, F16 or F20 (based on patients physical status) sterile plastic tube will be implemented at the level 4th or 5th intercostal space through the midaxillary line. However, in needle aspiration group, patients will be positioned semi-supine. Subsequently, G16 intravenous angiocath will be inserted through the midclavicular line at the level 2nd or 3rd intercostal space. The catheter needle will be removed and catheter will be fixed using sterile sticks. A three-way valve will be connected to the external end of the catheter and a 50 ml syringe will be connected to the valve. The air suction will be performed using 50 ml syringe till end of the air suction or up to 3.5 liters of air suctioning.

Hypothesis of present trial are as follows: a) repetitive needle aspiration may lead to higher treatment success rate in patients with primary spontaneous pneumothorax, in comparison to chest tube drainage, b) needle aspiration may result in reduction of hospital admission duration in patients with primary spontaneous pneumothorax compared to chest tube drainage, c) the rate of spontaneous pneumothorax recurrence during one-year follow-up might be lower in patients who undergo needle aspiration instead of chest tube drainage.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old
* Symptomatic primary spontaneous pneumothorax or intervention-needed spontaneous pneumothorax (pneumothorax more than 20% in volume due to Light criteria)

Exclusion Criteria:

* Tension pneumothorax
* bilateral severe respiratory failure
* demand for mechanical ventilation
* bilateral pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-08-12 (Actual); Primary Completion 2018-07-12 (Estimated); Study Completion 2018-10-12 (Estimated)

PRIMARY OUTCOMES:
Pneumothorax recurrence during one-year | One year postoperative
  Will be defined as the rate of pneumothorax recurrence until postoperative one-year.

SECONDARY OUTCOMES:
Successful treatment rate | Postoperative day 1 and postoperative day 7
  Is defined as completely resolved pneumothorax during admission.
Length of hospital admission | Through hospital admission, an average of 10 days
  will be calculated from the time of the operation to time of discharge.
Operation time | During procedure
  Will be calculated from the time of skin incision to completing the procedure including complete chest tube insertion in chest tube group or complete air suction or up to 3.5 liters of air suction in needle aspiration group.
Procedure induced complications | Postoperative day 1, Postoperative day 3, Postoperative day 7, Postoperative month 1,
  Includes all complications occurred during or after procedure during hospital stay.
Pneumothorax size | Before procedure, 1 hour after procedure, 48 hours after procedure, one-week after procedure
  Will be calculated by Light's formula using chest radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Reza hospital, Tabriz, East Azerbaijan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tschopp JM, Marquette CH. Spontaneous pneumothorax: stop chest tube as first-line therapy. Eur Respir J. 2017 Apr 12;49(4):1700306. doi: 10.1183/13993003.00306-2017. Print 2017 Apr. No abstract available. PMID 28404655
- [Background] Hu X, Cowl CT, Baqir M, Ryu JH. Air travel and pneumothorax. Chest. 2014 Apr;145(4):688-694. doi: 10.1378/chest.13-2363. PMID 24687705
- [Background] Cran IR, Rumball CA. Survey of spontaneous pneumothoraces in the Royal Air Force. Thorax. 1967 Sep;22(5):462-5. doi: 10.1136/thx.22.5.462. PMID 6050294
- [Background] Harvey J, Prescott RJ. Simple aspiration versus intercostal tube drainage for spontaneous pneumothorax in patients with normal lungs. British Thoracic Society Research Committee. BMJ. 1994 Nov 19;309(6965):1338-9. doi: 10.1136/bmj.309.6965.1338. No abstract available. PMID 7755720
- [Background] Dzeljilji A, Rokicki W, Rokicki M, Karus K. New aspects in the diagnosis and treatment of primary spontaneous pneumothorax. Kardiochir Torakochirurgia Pol. 2017 Mar;14(1):27-31. doi: 10.5114/kitp.2017.66926. Epub 2017 Mar 31. PMID 28515745
- [Background] MacDuff A, Arnold A, Harvey J; BTS Pleural Disease Guideline Group. Management of spontaneous pneumothorax: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii18-31. doi: 10.1136/thx.2010.136986. No abstract available. PMID 20696690
- [Background] Thelle A, Gjerdevik M, SueChu M, Hagen OM, Bakke P. Randomised comparison of needle aspiration and chest tube drainage in spontaneous pneumothorax. Eur Respir J. 2017 Apr 12;49(4):1601296. doi: 10.1183/13993003.01296-2016. Print 2017 Apr. PMID 28404647
- [Background] Tschopp JM, Bintcliffe O, Astoul P, Canalis E, Driesen P, Janssen J, Krasnik M, Maskell N, Van Schil P, Tonia T, Waller DA, Marquette CH, Cardillo G. ERS task force statement: diagnosis and treatment of primary spontaneous pneumothorax. Eur Respir J. 2015 Aug;46(2):321-35. doi: 10.1183/09031936.00219214. Epub 2015 Jun 25. PMID 26113675
- [Background] Wakai A, O'Sullivan RG, McCabe G. Simple aspiration versus intercostal tube drainage for primary spontaneous pneumothorax in adults. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD004479. doi: 10.1002/14651858.CD004479.pub2. PMID 17253510